CLINICAL TRIAL: NCT03233802
Title: Individualized Assessment and Treatment for Alcoholism: Treatment and Mechanisms
Brief Title: Individualized Assessment and Treatment for Alcoholism II
Acronym: IATP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Mark Litt, Professor of Behavioral Sciences, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-211-3; 1R01AA024729-01A1 (NIH)
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Alcoholism
Keywords: Alcohol Use Disorder; Treatment; Cognitive-Behavioral Treatment; Individualized Treatment
MeSH Terms: conditions — Alcoholism | interventions — Therapeutics; Case Management

STUDY DESIGN:
Intervention Model Description: 3 Group randomized clinical trial with parallel treatments
Who Masked: Investigator
Masking Description: Investigators are blind to treatment conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Individualized Assess & Treatment (IATP) (Experimental): Intervention: Cognitive-Behavioral IATP consists of 12 weekly visits of individual treatment. IATP employs cellphone-based experience sampling via interactive voice response (IVR) to assess drinking, plus craving, thoughts, feelings, and coping behaviors to develop near a real-time picture of patients' high-risk situations and the ways they use to deal with them. This information will be used by the therapist and client together to problem-solve and devise adaptive coping responses to these specific high-risk situations, and develop generalized solutions to deal with other situations in the future.
  Interventions: Behavioral: Individualized Assess & Treatment (IATP)
- Packaged Cognitive-Behavioral (PCBT) (Active Comparator): Intervention: Cognitive-Behavioral PCBT consists of 12 weekly visits of individual treatment. PCBT is designed to remediate deficits in skills for coping with interpersonal (e.g., social pressure, conflict with others) and intrapersonal (e.g., craving, anger) antecedents to drinking. The treatment consists of 6 mandatory modules (e.g., managing cravings) plus 6 electives from a list of 10 (e.g., receiving criticism; scheduling pleasant activities).The treatment, based on manuals developed for our previous clinical research provides a structured experience using didactic presentations, behavioral rehearsal, and homework practice exercises.
  Interventions: Behavioral: Packaged Cognitive-Behavioral (PCBT)
- Case Management (CaseM) (Active Comparator): Intervention: Social and Instrumental Support CaseM is included to control for cohort and other common factors in treatment. During the 12 individual CaseM sessions the therapist and participant will identify problems in daily living that may be of concern, and consider community resources that might help in dealing with them (e.g., contacting a psychiatrist for depression, or finding a better place to live). The therapist's role is to explore the patient's concerns, help to identify goals and resources, provide verbal support, and troubleshoot difficulties that may arise in obtaining or following through with services. The support and attention to ancillary services has proven effective in reducing drinking in previous studies.
  Interventions: Behavioral: Case Management (CaseM)

INTERVENTIONS:
Behavioral: Individualized Assess & Treatment (IATP) — See previous description
  Arms: Individualized Assess & Treatment (IATP)
Behavioral: Packaged Cognitive-Behavioral (PCBT) — See previous description
  Arms: Packaged Cognitive-Behavioral (PCBT)
Behavioral: Case Management (CaseM) — See previous description
  Arms: Case Management (CaseM)

SUMMARY:
The object of this study is to develop a treatment for alcohol use disorders that is more effective than current CB treatments. Through a 2009 R-21 pilot project the investigators developed a cognitive-behavioral (CB) treatment that employed cellphone-based experience sampling (ES) to collect detailed patient data, in near real-time, and that used those data to direct treatment for each patient based on his/her pattern of drinking and specific coping actions during high-risk situations. ES data included momentary assessments of situations, thoughts and feelings antecedent to drinking episodes, and the use of coping skills. That initial study of the Individualized Assessment and Treatment Program (IATP) showed promise. The present study is intended to extend the earlier findings, to compare IATP to a more active control treatment, and to evaluate long-term outcomes.

DETAILED DESCRIPTION:
An 2009 R-21 pilot project developed a cognitive-behavioral treatment for alcohol use disorders that employs cellphone-based experience sampling (ES) to collect detailed patient data in near real-time, and uses those data to direct treatment for each patient based on his/her specific patterns of drinking and specific coping actions during actual high-risk situations. ES data included situations, thoughts and feelings antecedent to drinking episodes, and any use of coping skills. The object was to create a CB treatment that was more relevant for each patient and more effective than current treatments. In the initial study the Individualized Assessment and Treatment Program (IATP) yielded better drinking rates at posttreatment, and more adaptive changes in coping, than a conventional manualized CBT program. Moreover, changes in drinking were partly mediated by pre-to-posttreatment changes in coping with high-risk situations. Questions unanswered included:

1. Because the pilot study only collected data pre- and posttreatment, with no follow-ups, it is not clear whether use of coping skills reduced drinking, or whether reduced drinking led to more adaptive coping.
2. It was not known which coping skills or other factors drive outcomes in the long-term.

To answer these and other questions the investigators proposed to enroll 207 patients in a full-scale trial of IATP with extended follow-ups to examine determinants of outcomes over time. IATP will be compared to a more conventional packaged CB treatment (PCBT), and to a Case Management Control condition (CaseM), in a dismantling design. In addition to coping, a number of other possible treatment mechanisms suggested by the literature will be examined, including motivation, self-efficacy, self-control, social support, alliance with the therapist, AA involvement, mindfulness, and utilization of other treatment services.

By specifically training coping skills for use in high-risk for drinking situations, the investigators will be able to assess how skills per se contribute to initiation and long-term maintenance of behavior change. The use of ES during treatment will allow a determination of what patients are actually doing, in close to real time, to initiate and maintain their own sobriety. The use of ES in the follow-up period will allow the investigators to determine whether coping skills that were active in initiation of reduced drinking continue to be active in the long-term, as well as the extent to which other mechanisms may come into play. In this way investigators can develop a clearer picture of the processes that affect outcomes of CBT, and will enable clinicians to focus more precisely on the most relevant mechanisms of change. Comparing IATP with PCBT will test effects of tailoring skills. The use of CaseM will control for the general effects of study participation (i.e., "common factors"), especially therapist support. The study builds on pilot data and on procedures that have already been developed but not fully tested. This would be the first study to evaluate effects of treatment on actual behaviors and cognitions in high-risk situations as they occur.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years old,
* Meet DSM-V criteria for Alcohol Use Disorder moderate-severe
* Willing to accept random assignment to any of the three conditions

Exclusion Criteria:

* Acute medical or psychiatric problems that require inpatient treatment (e.g., acute psychosis, or suicide/homicide risk)
* Reading ability below the fifth grade level
* Lack of reliable transportation to the treatment site, or excessive commuting distance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Proportion of days abstinent (PDA) | Every 3 months from intake through 21 months
  Proportion of days abstinent in the 90 days prior to each follow-up point

SECONDARY OUTCOMES:
Proportion Heavy Drinking days (PDH) | Every 3 months from intake through 21 months
  Proportion of days in which heavy drinking occurred in the 90 days prior to each follow-up point
Drinker Inventory of Consequences (DrInC) score | Every 6 months from intake through 21 months
  Negative life consequences of drinking

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Litt, Principal Investigator — UConn Health
Locations (1):
- UConn Health, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Litt MD, Tennen H, Kadden RM. Individualized Assessment and Treatment Program (IATP) for alcohol use disorder: Comparison with conventional cognitive-behavioral treatment and examination of coping skills as a mediator of treatment. J Consult Clin Psychol. 2024 Oct;92(10):711-726. doi: 10.1037/ccp0000907. Epub 2024 Oct 7. PMID 39374130